CLINICAL TRIAL: NCT04706676
Title: Integrative Neuromuscular Training in Adolescents and Children Treated for Cancer- a Multicenter Randomized Controlled Trial
Brief Title: Integrative Neuromuscular Training in Adolescents and Children Treated for Cancer
Acronym: INTERACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Hanne Baekgaard Larsen, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INTERACT-2020; 2019-5954 (Other Grant/Funding Number: The Children's Cancer Foundation); E-22597-01 (Other Grant/Funding Number: the Research Fund of Copenhagen University Hospital); 20-B-0409 (Other Grant/Funding Number: Helsefonden)
Record Dates: First submitted 2021-01-05; First posted 2021-01-13 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Cancer; Leukemia; Neoplasms; Lymphoma; Solid Tumor; CNS Tumor
Keywords: Pediatric Exercise Oncology; Integrative Neuromuscular Training; Children and Adolescents; ResistanceTraining; Metabolic Syndrome; Physical Activity; Motivation
MeSH Terms: conditions — Neoplasms; Leukemia; Lymphoma; Central Nervous System Neoplasms; Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrative neuromuscular training + motivational counseling + usual care (Experimental): General and specific strength and conditioning elements such as strength, power, motor skill training, dynamic stability, core-focused strength, plyometric and agility.
  Interventions: Behavioral: Integrative neuromuscular training (INT); Behavioral: motivational counseling session
- Active control group + motivational counseling + usual care (Active Comparator): home-based training program
  Interventions: Behavioral: Active control group: home-based training program; Behavioral: motivational counseling session

INTERVENTIONS:
Behavioral: Integrative neuromuscular training (INT) — Integrative neuromuscular training (INT), contains a multifaceted range of developmentally appropriate activities that incorporate general and specific strength and conditioning elements such as strength, power, motor skill training, dynamic stability, core-focused strength, plyometric and agility. INT can be camouflaged as games and play or performed as structured strength and conditioning program, depending on the participant's age, motor skill level and diagnosis. The intervention is designed to enhance health- and skill-related components of physical fitness.
  Parents or guardians will receive education in conducting INT at home, alongside an exercise-kit consisting of training equipment corresponding to the child's age and fitness level (fitness ropes, medicine ball, dumbbells).
  The INT group will receive usual standardized hospital care, including physiotherapy if needed.
  Arms: Integrative neuromuscular training + motivational counseling + usual care
Behavioral: Active control group: home-based training program — The active control group is offered a home-based training program consisting of combined aerobic, strength and stretching exercises. Further, they will receive monthly motivational consultations, as described below, concerning the training program. The use of the home-based training program will be monitored through exercise journals.
  The INT group will receive usual standardized hospital care, including physiotherapy if needed.
  Arms: Active control group + motivational counseling + usual care
Behavioral: motivational counseling session — Each child and their parents will participate in a monthly 30-minute motivational counseling session to adjust the intervention and training program according to the child's physical capacity and preferences. Further, the session will determine potential barriers towards performing physical exercise using the Self-efficacy for Exercise Scale.
  The sessions are based on the principles in Self-Determination Theory that includes a spectrum of external and internal motivation factors for engaging in exercise. Each session will provide guidelines to increase the general activity levels and adjust the intervention according to the child's preferences and presence of symptoms.

SUMMARY:
The INTERACT study is a nation-wide, population-based randomized controlled trial to investigate the effects of 6-month integrative neuromuscular training during anti-cancer treatment on lower body muscle strength, metabolic syndrome, various measures of physical function, physical activity, days of hospitalization, health-related quality of life and health behavior in children and adolescents with cancer. The increased insight derived from this study will impact the development of pediatric exercise oncology and be of high relevance to a broad group of children and adolescents with severe chronic illness.

The study is based on the overarching hypothesis, that structured integrative neuromuscular training initiated immediately after diagnosis will be effective in preventing deficits in neuromuscular function, limit long-term cardio-metabolic morbidity and found long-standing improvements in physical activity behavior.

To maintain adherence and motivation throughout a 6-month training intervention, weekly supervision of the training is needed. For this study, it is hypothesized that a supervised exercise intervention, in addition to a motivational counseling intervention and usual care, will improve muscle strength compared with unsupervised home-based training (active controls).

DETAILED DESCRIPTION:
Improved childhood cancer survival rates call for novel strategies to reduce acute and long-term physical complications of anti-cancer treatment.

Children with cancer have markedly impaired muscle strength, cardiorespiratory fitness, and physical function occurring few days after diagnosis - further declining because of anti-cancer treatment and physical inactivity during the treatment trajectory. Moreover, these impairments persist years after ended treatment. Further, the children become physically illiterate, which include a lack of confidence, competence and motivation to engage in physical activities. The combination of persistent physical complications and physical illiteracy predispose for metabolic- as well as musculoskeletal dysfunction that lead to severe medical conditions such as metabolic syndrome, diabetes and cardiovascular disease with reduced life-expectancy.

Studies indicate that structured exercise aimed to optimize both muscle and neuronal functions ('integrative neuromuscular training'), should be explored further to effectively counteract the impairment in physical function caused by childhood cancer and its treatment and found a more healthy lifestyle after ended treatment. This age-adjusted, strength-based exercise concept, based on games and play, is hypothesized to improve physical function in children and adolescents diagnosed with cancer.

The primary objective of this study is to investigate the effects of a 6-months integrative neuromuscular training intervention on knee extension strength in children and adolescents, ages 6-18 years, with cancer during anti-cancer treatment, compared with an active control group. Our secondary objectives are to investigate the effects of the intervention on markers of metabolic syndrome, hospitalized days, health-related quality of life, upper body muscle strength, cardiorespiratory fitness, physical function, physical activity behavior and body composition.

All outcomes, except hospitalized days, will be measured within 2 weeks of treatment initiation, 3-months after inclusion, after 6-months after inclusion, one month after ended treatment and 1 year after ended treatment.

The primary endpoint for the primary objective and secondary objectives, besides metabolic syndrome, are 6 months after treatment initiation. The primary endpoint for markers of metabolic syndrome will be 1 year after cessation of treatment

The INTERACT study is a national multicenter, two arm parallel group, randomized controlled superiority trial with 12 months follow-up after ended treatment, based in all national centers for pediatric oncology: University Hospital of Copenhagen (Rigshospitalet), Aarhus University Hospital and Odense University Hospital.

The study will include 127 children aged 6-18 years with any type of cancer that will be randomized (2:2) to either the intervention group (integrative neuromuscular training + motivational-counseling sessions + usual care) or active control group (home-based training program + motivational-counseling sessions + usual care) and stratified by sex, pubertal stage and diagnosis as 1) treatment for extracranial solid tumors and CNS-tumors; 2) treatment for hematologic malignancy 3) stem cell transplantation, within each hospital.

This intervention, integrative neuromuscular training (INT), contains a multifaceted range of developmentally appropriate activities that incorporate general and specific strength and conditioning elements such as strength, power, motor skill training, dynamic stability, core-focused strength, plyometric and agility. INT can be camouflaged as games and play or performed as structured strength and conditioning program, depending on the participant's age, motor skill level and diagnosis. The intervention is designed to enhance health- and skill-related components of physical fitness.

The integrative neuromuscular training group will in addition to usual care receive the intervention for six months.

All participants are recommended to participate in a minimum of 2 training session per week the first 7 weeks, and a minimum of three session per week from week 8-24. During the intense phase of treatment (first six months of treatment), all participants indifferent of cancer type will receive combinations of treatment requiring either hospitalization or visits to the outpatient clinic at least once per week. The participants, therefore, receives supervised training at least once per week. All other training session is conducted as home-based training. If there are weeks, without any visits to the hospital or outpatient clinic, all training session will be conducted at home. In this case, the participants will receive a phone call from the intervention physiotherapist concerning questions, exercise choice and intensity of exercises.

Parents or guardians will receive education in conducting INT at home, alongside an exercise-kit consisting of training equipment corresponding to the child's age and fitness level (fitness ropes, medicine ball, dumbbells).

The active control group is, in addition to usual care, offered a home-based training program consisting of combined aerobic, strength and stretching exercises.

Participants in both groups will receive a monthly 30-minute motivational-counseling session to adjust the intervention and training program according to the child's physical capacity and preferences. Further, the session will determine potential barriers towards performing physical exercise using the Self-efficacy for Exercise Scale.

Both groups receive standardized hospital care, usual care, including physiotherapy if needed

Sample size:

A difference of 10 % as a result of physical exercise is regarded as a clinically relevant change (1). Based on a mean 41.4 +/- 7.6 (2) and a 10% increase, an alpha level of 0.05 and power of 80%, 106 children are needed. Approximately, 60 children with cancer at the age of 6-18 years will be diagnosed pr. year at Copenhagen University Hospital, Rigshospitalet Aarhus University Hospital and Odense University Hospital. Assuming a 20 % dropout rate, a total of 2.2 years is needed to include the required number of children with cancer (n=127).

A blinded statistician will randomize participants to either intervention or active control group using a computer-generated concealed allocation procedure, to secure a proportionate stratified random sample.

Due to the nature of the intervention, neither participants, nor assessors, will be blinded to the allocation.

ELIGIBILITY:
Inclusion Criteria:

* All malign and benign disorders treated with chemotherapy and/or irradiation

Exclusion Criteria:

* Severe mental and/or physical disability, i.e. participants where all types of physical training and testing of physical function are contraindicated
* terminal illness
* unable to communicate in Danish

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Lower extremity isometric knee extension strength | Within 2 weeks of treatment initiation (baseline)
  Isometric leg extension is tested using a special-build strength ergometer (Gym 2000®) with a dynamometer (US2A100 kg, Holtinger, Germany).
  The participant is instructed to kick (forward) with maximal force keeping maximal intensity for at least five seconds. Three attempts with a two minutes break is carried out, however the participant can try as many attempts as possible if the participant keeps showing improvements. Highest score is noted.
  The participant is sitting upright with hands grasping the bench. Hips and knees are kept in 90 degrees flexion. The height of the bench is adjusted to maintain both feet of the ground.
  The chain to the dynamometer is adjusted in order to keep the leg in 90 degrees flexion during muscle contraction. The test is performed unilaterally, and in some cases solely on one leg as children with solid tumors in under extremities may be restricted to testing.
Lower extremity isometric knee extension strength | 3-months after inclusion
  Isometric leg extension is tested using a special-build strength ergometer (Gym 2000®) with a dynamometer (US2A100 kg, Holtinger, Germany).
  The participant is instructed to kick (forward) with maximal force keeping maximal intensity for at least five seconds. Three attempts with a two minutes break is carried out, however the participant can try as many attempts as possible if the participant keeps showing improvements. Highest score is noted.
  The participant is sitting upright with hands grasping the bench. Hips and knees are kept in 90 degrees flexion. The height of the bench is adjusted to maintain both feet of the ground.
  The chain to the dynamometer is adjusted in order to keep the leg in 90 degrees flexion during muscle contraction. The test is performed unilaterally, and in some cases solely on one leg as children with solid tumors in under extremities may be restricted to testing.
Lower extremity isometric knee extension strength | 6-months after inclusion (primary endpoint)
  Isometric leg extension is tested using a special-build strength ergometer (Gym 2000®) with a dynamometer (US2A100 kg, Holtinger, Germany).
  The participant is instructed to kick (forward) with maximal force keeping maximal intensity for at least five seconds. Three attempts with a two minutes break is carried out, however the participant can try as many attempts as possible if the participant keeps showing improvements. Highest score is noted.
  The participant is sitting upright with hands grasping the bench. Hips and knees are kept in 90 degrees flexion. The height of the bench is adjusted to maintain both feet of the ground.
  The chain to the dynamometer is adjusted in order to keep the leg in 90 degrees flexion during muscle contraction. The test is performed unilaterally, and in some cases solely on one leg as children with solid tumors in under extremities may be restricted to testing.
Lower extremity isometric knee extension strength | 1 month after ended treatment
  Isometric leg extension is tested using a special-build strength ergometer (Gym 2000®) with a dynamometer (US2A100 kg, Holtinger, Germany).
  The participant is instructed to kick (forward) with maximal force keeping maximal intensity for at least five seconds. Three attempts with a two minutes break is carried out, however the participant can try as many attempts as possible if the participant keeps showing improvements. Highest score is noted.
  The participant is sitting upright with hands grasping the bench. Hips and knees are kept in 90 degrees flexion. The height of the bench is adjusted to maintain both feet of the ground.
  The chain to the dynamometer is adjusted in order to keep the leg in 90 degrees flexion during muscle contraction. The test is performed unilaterally, and in some cases solely on one leg as children with solid tumors in under extremities may be restricted to testing.
Lower extremity isometric knee extension strength | 1 year after ended treatment
  Isometric leg extension is tested using a special-build strength ergometer (Gym 2000®) with a dynamometer (US2A100 kg, Holtinger, Germany).
  The participant is instructed to kick (forward) with maximal force keeping maximal intensity for at least five seconds. Three attempts with a two minutes break is carried out, however the participant can try as many attempts as possible if the participant keeps showing improvements. Highest score is noted.
  The participant is sitting upright with hands grasping the bench. Hips and knees are kept in 90 degrees flexion. The height of the bench is adjusted to maintain both feet of the ground.
  The chain to the dynamometer is adjusted in order to keep the leg in 90 degrees flexion during muscle contraction. The test is performed unilaterally, and in some cases solely on one leg as children with solid tumors in under extremities may be restricted to testing.

SECONDARY OUTCOMES:
Markers of metabolic syndrome: Waist circumference (primary secondary outcome) | within 2 weeks of treatment initiation
  Waist circumference is measured in CM, at the end of several consecutive natural breaths, at a level parallel to the floor, midpoint between the top of the iliac crest and the lower margin of the last palpable rib in the mid axillary line following standards described by the World Health Organization. Metabolic syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: triglycerides (primary secondary outcome) | within 2 weeks of treatment initiation
  Blood samples will be drawn from an antecubital vein, or when possible, through a central or peripheral venous catheter. Markers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: high-density lipoprotein (HDL) cholesterol (primary secondary outcome) | within 2 weeks of treatment initiation
  Blood samples will be drawn from an antecubital vein, or when possible, through a central or peripheral venous catheter. Markers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: blood pressure (primary secondary outcome) | within 2 weeks of treatment initiation
  Blood pressure (mmHg) will be measured in the morning and in the right arm with the subject in the sitting position. TMarkers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: fasting blood sugar and insulin (primary secondary outcome) | within 2 weeks of treatment initiation
  Blood samples will be drawn from an antecubital vein, or when possible, through a central or peripheral venous catheter. Markers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: Waist circumference (primary secondary outcome) | 6 months after inclusion (before a treatment block)
  Waist circumference is measured in CM, at the end of several consecutive natural breaths, at a level parallel to the floor, midpoint between the top of the iliac crest and the lower margin of the last palpable rib in the mid axillary line following standards described by the World Health Organization. Metabolic syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: triglycerides (primary secondary outcome) | 6 months after inclusion (before a treatment block)
  Blood samples will be drawn from an antecubital vein, or when possible, through a central or peripheral venous catheter. Markers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: high-density lipoprotein (HDL) cholesterol (primary secondary outcome) | 6 months after inclusion (before a treatment block)
  Blood samples will be drawn from an antecubital vein, or when possible, through a central or peripheral venous catheter. Markers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: blood pressure (primary secondary outcome) | 6 months after inclusion (before a treatment block)
  Blood samples will be drawn from an antecubital vein, or when possible, through a central or peripheral venous catheter. Markers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: fasting blood sugar and insulin (primary secondary outcome) | 6 months after inclusion (before a treatment block)
  Blood samples will be drawn from an antecubital vein, or when possible, through a central or peripheral venous catheter. Markers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: Waist circumference (primary secondary outcome) | 1 month after ended treatment
  Waist circumference is measured in CM, at the end of several consecutive natural breaths, at a level parallel to the floor, midpoint between the top of the iliac crest and the lower margin of the last palpable rib in the mid axillary line following standards described by the World Health Organization. Metabolic syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: triglycerides (primary secondary outcome) | 1 month after ended treatment
  Blood samples will be drawn from an antecubital vein, or when possible, through a central or peripheral venous catheter. Markers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: high-density lipoprotein (HDL) cholesterol(primary secondary outcome) | 1 month after ended treatment
  Blood samples will be drawn from an antecubital vein, or when possible, through a central or peripheral venous catheter. Markers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: blood pressure (primary secondary outcome) | 1 month after ended treatment
  Blood samples will be drawn from an antecubital vein, or when possible, through a central or peripheral venous catheter. Markers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: fasting blood sugar and insulin (primary secondary outcome) | 1 month after ended treatment
  Blood samples will be drawn from an antecubital vein, or when possible, through a central or peripheral venous catheter. Markers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: Waist circumference (primary secondary outcome) | 1 year after end of treatment (primary endpoint)
  Waist circumference is measured in CM, at the end of several consecutive natural breaths, at a level parallel to the floor, midpoint between the top of the iliac crest and the lower margin of the last palpable rib in the mid axillary line following standards described by the World Health Organization. Metabolic syndrome is based on age-based criterias defined by the International Diabetes Foundation (3.
Markers of metabolic syndrome: triglycerides (primary secondary outcome) | 1 year after end of treatment (primary endpoint)
  Blood samples will be drawn from an antecubital vein, or when possible, through a central or peripheral venous catheter. Markers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: high-density lipoprotein (HDL) cholesterol (primary secondary outcome) | 1 year after end of treatment (primary endpoint)
  Blood samples will be drawn from an antecubital vein, or when possible, through a central or peripheral venous catheter. Markers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: blood pressure (primary secondary outcome) | 1 year after end of treatment (primary endpoint)
  Blood samples will be drawn from an antecubital vein, or when possible, through a central or peripheral venous catheter. Markers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Markers of metabolic syndrome: fasting blood sugar and insulin (primary secondary outcome) | 1 year after end of treatment (primary endpoint)
  Blood samples will be drawn from an antecubital vein, or when possible, through a central or peripheral venous catheter. Markers of Metabolic Syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Isometric Bench Press | Within 2 weeks of treatment initiation (baseline)
  Isometric bench press is tested using a special-build strength ergometer (Gym 2000®) with a dynamometer (US2A100 kg, Holtinger, Germany).
  The participant lies in supine position, with shoulder in 150% of biacromial width and elbows in 90 degrees flexion, with the height of the bar adjusted accordingly. The participant is obliged to maintain this position during the test. The participant is instructed to push (upwards) with maximal force.
Isometric Bench Press | 3-months after inclusion
  Isometric bench press is tested using a special-build strength ergometer (Gym 2000®) with a dynamometer (US2A100 kg, Holtinger, Germany).
  The participant lies in supine position, with shoulder in 150% of biacromial width and elbows in 90 degrees flexion, with the height of the bar adjusted accordingly. The participant is obliged to maintain this position during the test. The participant is instructed to push (upwards) with maximal force.
Isometric Bench Press | 6-months after inclusion (primary endpoint)
  Isometric bench press is tested using a special-build strength ergometer (Gym 2000®) with a dynamometer (US2A100 kg, Holtinger, Germany).
  The participant lies in supine position, with shoulder in 150% of biacromial width and elbows in 90 degrees flexion, with the height of the bar adjusted accordingly. The participant is obliged to maintain this position during the test. The participant is instructed to push (upwards) with maximal force.
Isometric Bench Press | 1 month after ended treatment
  Isometric bench press is tested using a special-build strength ergometer (Gym 2000®) with a dynamometer (US2A100 kg, Holtinger, Germany).
  The participant lies in supine position, with shoulder in 150% of biacromial width and elbows in 90 degrees flexion, with the height of the bar adjusted accordingly. The participant is obliged to maintain this position during the test. The participant is instructed to push (upwards) with maximal force.
Isometric Bench Press | 1 year after ended treatment
  Isometric bench press is tested using a special-build strength ergometer (Gym 2000®) with a dynamometer (US2A100 kg, Holtinger, Germany).
  The participant lies in supine position, with shoulder in 150% of biacromial width and elbows in 90 degrees flexion, with the height of the bar adjusted accordingly. The participant is obliged to maintain this position during the test. The participant is instructed to push (upwards) with maximal force.
Hand Grip strength | Within 2 weeks of treatment initiation (baseline)
  Handgrip strength is measured using a hand-held dynamometer. Participants are placed in a seated position with the elbow flexed at 90°, with three attempts performed for each hand. During testing, the participant will be encouraged to exhibit the best possible force, and the best measure in the strongest hand will be used as test score. Hand Grip strength is also used as a surrogate measure for upper-body physical function.
Hand Grip strength | 3-months after inclusion
  Handgrip strength is measured using a hand-held dynamometer. Participants are placed in a seated position with the elbow flexed at 90°, with three attempts performed for each hand. During testing, the participant will be encouraged to exhibit the best possible force, and the best measure in the strongest hand will be used as test score. Hand Grip strength is also used as a surrogate measure for upper-body physical function.
Hand Grip strength | 6-months after inclusion (primary endpoint)
  Handgrip strength is measured using a hand-held dynamometer. Participants are placed in a seated position with the elbow flexed at 90°, with three attempts performed for each hand. During testing, the participant will be encouraged to exhibit the best possible force, and the best measure in the strongest hand will be used as test score. Hand Grip strength is also used as a surrogate measure for upper-body physical function.
Hand Grip strength | 1 month after ended treatment
  Handgrip strength is measured using a hand-held dynamometer. Participants are placed in a seated position with the elbow flexed at 90°, with three attempts performed for each hand. During testing, the participant will be encouraged to exhibit the best possible force, and the best measure in the strongest hand will be used as test score. Hand Grip strength is also used as a surrogate measure for upper-body physical function.
Hand Grip strength | 1 year after ended treatment
  Handgrip strength is measured using a hand-held dynamometer. Participants are placed in a seated position with the elbow flexed at 90°, with three attempts performed for each hand. During testing, the participant will be encouraged to exhibit the best possible force, and the best measure in the strongest hand will be used as test score. Hand Grip strength is also used as a surrogate measure for upper-body physical function.
Six Minutes Walk Test | Within 2 weeks of treatment initiation (baseline)
  Maximal walking distance in six minutes, as a surrogate measure for cardiorespiratory fitness, is measured through the self-paced 6-minute walk test. Two cones are positioned on a straight course spaced at 20 m. The object of the test is to walk as far as possible in 6 minutes. Participants must walk back and forth around the cones, permitted to slow down, to stop, and to rest as necessary without running or jogging. The accumulated distance is noted, and degree of perceived exhaustion is estimated using the Borg Category-Ratio 1-10 Scale.
Six Minutes Walk Test | 3-months after inclusion
  Maximal walking distance in six minutes, as a surrogate measure for cardiorespiratory fitness, is measured through the self-paced 6-minute walk test. Two cones are positioned on a straight course spaced at 20 m. The object of the test is to walk as far as possible in 6 minutes. Participants must walk back and forth around the cones, permitted to slow down, to stop, and to rest as necessary without running or jogging. The accumulated distance is noted, and degree of perceived exhaustion is estimated using the Borg Category-Ratio 1-10 Scale.
Six Minutes Walk Test | 6-months after inclusion (primary endpoint)
  Maximal walking distance in six minutes, as a surrogate measure for cardiorespiratory fitness, is measured through the self-paced 6-minute walk test. Two cones are positioned on a straight course spaced at 20 m. The object of the test is to walk as far as possible in 6 minutes. Participants must walk back and forth around the cones, permitted to slow down, to stop, and to rest as necessary without running or jogging. The accumulated distance is noted, and degree of perceived exhaustion is estimated using the Borg Category-Ratio 1-10 Scale.
Six Minutes Walk Test | 1 month after ended treatment
  Maximal walking distance in six minutes, as a surrogate measure for cardiorespiratory fitness, is measured through the self-paced 6-minute walk test. Two cones are positioned on a straight course spaced at 20 m. The object of the test is to walk as far as possible in 6 minutes. Participants must walk back and forth around the cones, permitted to slow down, to stop, and to rest as necessary without running or jogging. The accumulated distance is noted, and degree of perceived exhaustion is estimated using the Borg Category-Ratio 1-10 Scale.
Six Minutes Walk Test | 1 year after ended treatment
  Maximal walking distance in six minutes, as a surrogate measure for cardiorespiratory fitness, is measured through the self-paced 6-minute walk test. Two cones are positioned on a straight course spaced at 20 m. The object of the test is to walk as far as possible in 6 minutes. Participants must walk back and forth around the cones, permitted to slow down, to stop, and to rest as necessary without running or jogging. The accumulated distance is noted, and degree of perceived exhaustion is estimated using the Borg Category-Ratio 1-10 Scale.
Thirty Seconds and One-Minute Sit-to-stand | Within 2 weeks of treatment initiation (baseline)
  Sit-To-Stand is performed using a chair that allows the child to flex the legs at a 90o angle. The child is instructed to fold his/her arms across the chest or to let them hang to the side, stand straight and then touch the chair with their bottom while returning to a seated position. Strong verbal encouragement will be given during the test. Subjects were permitted to use rest periods to complete the one-minute period. The test score equates the number of repetitions during a 60 second period. As a marker for lower extremity muscle strength, the number repetition completed after 30 seconds will be noted.
Thirty Seconds and One-Minute Sit-to-stand | 3-months after inclusion
  Sit-To-Stand is performed using a chair that allows the child to flex the legs at a 90o angle. The child is instructed to fold his/her arms across the chest or to let them hang to the side, stand straight and then touch the chair with their bottom while returning to a seated position. Strong verbal encouragement will be given during the test. Subjects were permitted to use rest periods to complete the one-minute period. The test score equates the number of repetitions during a 60 second period. As a marker for lower extremity muscle strength, the number repetition completed after 30 seconds will be noted.
Thirty Seconds and One-Minute Sit-to-stand | 6-months after inclusion (primary endpoint)
  Sit-To-Stand is performed using a chair that allows the child to flex the legs at a 90o angle. The child is instructed to fold his/her arms across the chest or to let them hang to the side, stand straight and then touch the chair with their bottom while returning to a seated position. Strong verbal encouragement will be given during the test. Subjects were permitted to use rest periods to complete the one-minute period. The test score equates the number of repetitions during a 60 second period. As a marker for lower extremity muscle strength, the number repetition completed after 30 seconds will be noted.
The timed Up-and-Go Test: | 3-months after inclusion
  The timed Up-and-Go test (TUG) tests basic mobility, defined as the ability to get in and out of bed, to get up and down from a chair, to walk short distances, and to turn.
  The test is performed using a chair that allows the child to flex the legs at a 90o angle. From the start position, with the back resting against the chair and arms on knees, the child is instructed to stand up, walk three meters as fast as possible, turn around and return to the start position. Completion time will be recorded in seconds to the nearest two decimals. Strong verbal encouragement will be given during the test. The lowest score of three tries will be used in the analysis.
Thirty Seconds and One-Minute Sit-to-stand | 1 month after ended treatment
  Sit-To-Stand is performed using a chair that allows the child to flex the legs at a 90o angle. The child is instructed to fold his/her arms across the chest or to let them hang to the side, stand straight and then touch the chair with their bottom while returning to a seated position. Strong verbal encouragement will be given during the test. Subjects were permitted to use rest periods to complete the one-minute period. The test score equates the number of repetitions during a 60 second period. As a marker for lower extremity muscle strength, the number repetition completed after 30 seconds will be noted.
Thirty Seconds and One-Minute Sit-to-stand | 1 year after ended treatment
  Sit-To-Stand is performed using a chair that allows the child to flex the legs at a 90o angle. The child is instructed to fold his/her arms across the chest or to let them hang to the side, stand straight and then touch the chair with their bottom while returning to a seated position. Strong verbal encouragement will be given during the test. Subjects were permitted to use rest periods to complete the one-minute period. The test score equates the number of repetitions during a 60 second period. As a marker for lower extremity muscle strength, the number repetition completed after 30 seconds will be noted.
The timed Up-and-Go Test: | Within 2 weeks of treatment initiation (baseline)
  The timed Up-and-Go test (TUG) tests basic mobility, defined as the ability to get in and out of bed, to get up and down from a chair, to walk short distances, and to turn.
  The test is performed using a chair that allows the child to flex the legs at a 90o angle. From the start position, with the back resting against the chair and arms on knees, the child is instructed to stand up, walk three meters as fast as possible, turn around and return to the start position. Completion time will be recorded in seconds to the nearest two decimals. Strong verbal encouragement will be given during the test. The lowest score of three tries will be used in the analysis.
The timed Up-and-Go Test: | 6-months after inclusion (primary endpoint)
  The timed Up-and-Go test (TUG) tests basic mobility, defined as the ability to get in and out of bed, to get up and down from a chair, to walk short distances, and to turn.
  The test is performed using a chair that allows the child to flex the legs at a 90o angle. From the start position, with the back resting against the chair and arms on knees, the child is instructed to stand up, walk three meters as fast as possible, turn around and return to the start position. Completion time will be recorded in seconds to the nearest two decimals. Strong verbal encouragement will be given during the test. The lowest score of three tries will be used in the analysis.
The timed Up-and-Go Test: | 1 month after ended treatment
  The timed Up-and-Go test (TUG) tests basic mobility, defined as the ability to get in and out of bed, to get up and down from a chair, to walk short distances, and to turn.
  The test is performed using a chair that allows the child to flex the legs at a 90o angle. From the start position, with the back resting against the chair and arms on knees, the child is instructed to stand up, walk three meters as fast as possible, turn around and return to the start position. Completion time will be recorded in seconds to the nearest two decimals. Strong verbal encouragement will be given during the test. The lowest score of three tries will be used in the analysis.
The timed Up-and-Go Test: | 1 year after ended treatment
  The timed Up-and-Go test (TUG) tests basic mobility, defined as the ability to get in and out of bed, to get up and down from a chair, to walk short distances, and to turn.
  The test is performed using a chair that allows the child to flex the legs at a 90o angle. From the start position, with the back resting against the chair and arms on knees, the child is instructed to stand up, walk three meters as fast as possible, turn around and return to the start position. Completion time will be recorded in seconds to the nearest two decimals. Strong verbal encouragement will be given during the test. The lowest score of three tries will be used in the analysis.
Hospitalized days | measured 6 months after inclusion (primary endpoint)
  Number of admissions to hospital (total number of admissions, scheduled and unscheduled admission) will be drawn from the participants medical records
Hospitalized days | 1month after ended treatment
  Number of admissions to hospital (total number of admissions, scheduled and unscheduled admission) will be drawn from the participants medical records
Hospitalized days | 1 year after ended treatment
  Number of admissions to hospital (total number of admissions, scheduled and unscheduled admission) will be drawn from the participants medical records
Body composition: Bone Mineral Density | within 2 weeks of treatment initiation
  Bone Mineral Density (g/cm2) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Bone Mineral Content | within 2 weeks of treatment initiation
  Bone Mineral content (kg) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Body Fat | within 2 weeks of treatment initiation
  Body Fat (kg and %) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Fat-Free Mass | within 2 weeks of treatment initiation
  Fat-Free Mass (kg and %) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Bone Mineral Density | 6 months after inclusion (before a treatment block)
  Bone Mineral Density (g/cm2) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Bone Mineral Content | 6 months after inclusion (before a treatment block)
  Bone Mineral Content (kg) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Body Fat | 6 months after inclusion (before a treatment block)
  Body Fat (kg and %) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Fat-Free Mass | 6 months after inclusion (before a treatment block)
  Fat-Free Mass (kg and %) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Bone Mineral Density | 1 month after ended treatment.
  Bone Mineral Density (g/cm2) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Bone Mineral Content | 1 month after ended treatment.
  Bone Mineral Content (kg) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Body Fat | 1 month after ended treatment.
  Body Fat (kg and %) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Fat-Free Mass | 1 month after ended treatment.
  Fat-Free Mass (kg and %) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Bone Mineral Density | 1 year after end of treatment (primary endpoint).
  Bone Mineral Density (g/cm2) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Bone Mineral Content | 1 year after end of treatment (primary endpoint).
  Bone Mineral Content (kg) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Body Fat | 1 year after end of treatment (primary endpoint).
  Body Fat (kg and %) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Fat-Free Mass | 1 year after end of treatment (primary endpoint).
  Fat-Free Mass (kg and %) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
The PedsQL Generic Core Scale: Young Child, Children, Teens Self-Report and Parent Proxy-Report: | Within 2 weeks of treatment initiation
  The Pediatric Quality of Life Inventory (PedsQL Core) measures the quality of life in children using 23 items on a five-point response scale from never to almost always. The answers are divided into four domains: health and physical activity, emotions, dealing with others, and school activity.
The PedsQL Generic Core Scale: Young Child, Children, Teens Self-Report and Parent Proxy-Report: | 6-months after inclusion.
  The Pediatric Quality of Life Inventory (PedsQL Core) measures the quality of life in children using 23 items on a five-point response scale from never to almost always. The answers are divided into four domains: health and physical activity, emotions, dealing with others, and school activity.
The PedsQL Generic Core Scale: Young Child, Children, Teens Self-Report and Parent Proxy-Report: | 1 month after ended treatment
  The Pediatric Quality of Life Inventory (PedsQL Core) measures the quality of life in children using 23 items on a five-point response scale from never to almost always. The answers are divided into four domains: health and physical activity, emotions, dealing with others, and school activity.
The PedsQL Generic Core Scale: Young Child, Children, Teens Self-Report and Parent Proxy-Report: | 1 year after ended treatment
  The Pediatric Quality of Life Inventory (PedsQL Core) measures the quality of life in children using 23 items on a five-point response scale from never to almost always. The answers are divided into four domains: health and physical activity, emotions, dealing with others, and school activity.
Prevalence of metabolic syndrome | within 2 weeks of treatment initiation.
  Prevalence of Metabolic syndrome, based on markers described above (waist circumference, triglycerides, high-density lipoprotein (HDL) cholesterol, blood pressure, fasting blood sugar and insulin) will be calculated in the Intervention and active control group. Although Children between 6 and 9.9 years cannot be diagnosed with Metabolic syndrome, the potential decline or increase in the biological markers, i.e. predisposition, for metabolic syndrome will, however, be described in this study.
Prevalence of metabolic syndrome | 6 months after inclusion (before a treatment block)
  Prevalence of Metabolic syndrome, based on markers described above (waist circumference, triglycerides, high-density lipoprotein (HDL) cholesterol, blood pressure, fasting blood sugar and insulin) will be calculated in the Intervention and active control group. Although Children between 6 and 9.9 years cannot be diagnosed with Metabolic syndrome, the potential decline or increase in the biological markers, i.e. predisposition, for metabolic syndrome will, however, be described in this study.
Prevalence of metabolic syndrome | 1 month after ended treatment.
  Prevalence of Metabolic syndrome, based on markers described above (waist circumference, triglycerides, high-density lipoprotein (HDL) cholesterol, blood pressure, fasting blood sugar and insulin) will be calculated in the Intervention and active control group. Although Children between 6 and 9.9 years cannot be diagnosed with Metabolic syndrome, the potential decline or increase in the biological markers, i.e. predisposition, for metabolic syndrome will, however, be described in this study.
Prevalence of metabolic syndrome | 1 year after end of treatment (primary endpoint)
  Prevalence of Metabolic syndrome, based on markers described above (waist circumference, triglycerides, high-density lipoprotein (HDL) cholesterol, blood pressure, fasting blood sugar and insulin) will be calculated in the Intervention and active control group. Although Children between 6 and 9.9 years cannot be diagnosed with Metabolic syndrome, the potential decline or increase in the biological markers, i.e. predisposition, for metabolic syndrome will, however, be described in this study.

OTHER OUTCOMES:
Metabolomics (explorative outcome) | within 2 weeks of treatment initiation, at 6 months (before a treatment block), one month after ended treatment and 1 year after end of treatment.
  Metabolomics will be performed in urine and plasma for deep metabolomic phenotyping in collaboration with professor L.O. Dragsted (University of Copenhagen). The metabolites (<1500 Da) will be profiled by reversed-phase ultra-high-performance liquid chromatography coupled with a quadrupole - time-of-flight dual mass spectrometer.
Metabolomics (explorative outcome) | 6 months after inclusion (before a treatment block.
  Metabolomics will be performed in urine and plasma for deep metabolomic phenotyping in collaboration with professor L.O. Dragsted (University of Copenhagen). The metabolites (<1500 Da) will be profiled by reversed-phase ultra-high-performance liquid chromatography coupled with a quadrupole - time-of-flight dual mass spectrometer.
Metabolomics (explorative outcome) | 1 month after ended treatment.
  Metabolomics will be performed in urine and plasma for deep metabolomic phenotyping in collaboration with professor L.O. Dragsted (University of Copenhagen). The metabolites (<1500 Da) will be profiled by reversed-phase ultra-high-performance liquid chromatography coupled with a quadrupole - time-of-flight dual mass spectrometer.
Metabolomics (explorative outcome) | 1 year after end of treatment.
  Metabolomics will be performed in urine and plasma for deep metabolomic phenotyping in collaboration with professor L.O. Dragsted (University of Copenhagen). The metabolites (<1500 Da) will be profiled by reversed-phase ultra-high-performance liquid chromatography coupled with a quadrupole - time-of-flight dual mass spectrometer.
Dietary assessment (explorative outcome) | within 2 weeks of treatment initiation
  Collection of information regarding the participants dietary intake is based on self-reporting during 3-5days in the online diet program 'Madlog' (Madlog Vita, Vitakost, Kolding Denmark). An overall report of intake calculated in both macro and micronutrients is determined based on the Danish Technical University's (DTU) and the Danish Food Institute's database FRIDA (Frida.com)
Dietary assessment (explorative outcome) | 6 months after inclusion (before a treatment block),
  Collection of information regarding the participants dietary intake is based on self-reporting during 3-5days in the online diet program 'Madlog' (Madlog Vita, Vitakost, Kolding Denmark). An overall report of intake calculated in both macro and micronutrients is determined based on the Danish Technical University's (DTU) and the Danish Food Institute's database FRIDA (Frida.com)
Dietary assessment (explorative outcome) | 1 month after ended treatment.
  Collection of information regarding the participants dietary intake is based on self-reporting during 3-5days in the online diet program 'Madlog' (Madlog Vita, Vitakost, Kolding Denmark). An overall report of intake calculated in both macro and micronutrients is determined based on the Danish Technical University's (DTU) and the Danish Food Institute's database FRIDA (Frida.com)
Dietary assessment (explorative outcome) | 1 year after end of treatment.
  Collection of information regarding the participants dietary intake is based on self-reporting during 3-5days in the online diet program 'Madlog' (Madlog Vita, Vitakost, Kolding Denmark). An overall report of intake calculated in both macro and micronutrients is determined based on the Danish Technical University's (DTU) and the Danish Food Institute's database FRIDA (Frida.com)
Intestinal microbiota (explorative outcome) | within 2 weeks of treatment initiation, at 6 months (before a treatment block), one month after ended treatment and 1 year after end of treatment.
  Total DNA will be extracted from fecal samples using the Illumina HiSeq technology, generating16S data with the option to later run full microbiome sequencing on selected samples. These studies will be done in collaboration with the National Food Institute, Technical University of Denmark
Intestinal microbiota (explorative outcome) | within 2 weeks of treatment initiation.
  Total DNA will be extracted from fecal samples using the Illumina HiSeq technology, generating16S data with the option to later run full microbiome sequencing on selected samples. These studies will be done in collaboration with the National Food Institute, Technical University of Denmark
Intestinal microbiota (explorative outcome) | 6 months after inclusion (before a treatment block.
  Total DNA will be extracted from fecal samples using the Illumina HiSeq technology, generating16S data with the option to later run full microbiome sequencing on selected samples. These studies will be done in collaboration with the National Food Institute, Technical University of Denmark
Intestinal microbiota (explorative outcome) | 1month after ended treatment.
  Total DNA will be extracted from fecal samples using the Illumina HiSeq technology, generating16S data with the option to later run full microbiome sequencing on selected samples. These studies will be done in collaboration with the National Food Institute, Technical University of Denmark
Intestinal microbiota (explorative outcome) | 1 year after end of treatment.
  Total DNA will be extracted from fecal samples using the Illumina HiSeq technology, generating16S data with the option to later run full microbiome sequencing on selected samples. These studies will be done in collaboration with the National Food Institute, Technical University of Denmark
Inflammatory cytokines and mediators (explorative outcome) | within 2 weeks of treatment initiation
  Blood samples will be analyzed for inflammation-related growth factors, chemokines, incretins, epithelial and endothelial markers and cytokines including interleukin 6 (IL-6), tumor necrosis factor-alpha (TNF-α) and macrophage-related biomarkers (sCD163 and sCD206), by ELISA or by the Luminex at the Institute of Inflammation Research, Copenhagen University Hospital, Rigshospitalet.
Inflammatory cytokines and mediators (explorative outcome) | 6 months after inclusion (before a treatment block).
  Blood samples will be analyzed for inflammation-related growth factors, chemokines, incretins, epithelial and endothelial markers and cytokines including interleukin 6 (IL-6), tumor necrosis factor-alpha (TNF-α) and macrophage-related biomarkers (sCD163 and sCD206), by ELISA or by the Luminex at the Institute of Inflammation Research, Copenhagen University Hospital, Rigshospitalet.
Inflammatory cytokines and mediators (explorative outcome) | 1 month after ended treatment.
  Blood samples will be analyzed for inflammation-related growth factors, chemokines, incretins, epithelial and endothelial markers and cytokines including interleukin 6 (IL-6), tumor necrosis factor-alpha (TNF-α) and macrophage-related biomarkers (sCD163 and sCD206), by ELISA or by the Luminex at the Institute of Inflammation Research, Copenhagen University Hospital, Rigshospitalet.
Inflammatory cytokines and mediators (explorative outcome) | 1 year after end of treatment.
  Blood samples will be analyzed for inflammation-related growth factors, chemokines, incretins, epithelial and endothelial markers and cytokines including interleukin 6 (IL-6), tumor necrosis factor-alpha (TNF-α) and macrophage-related biomarkers (sCD163 and sCD206), by ELISA or by the Luminex at the Institute of Inflammation Research, Copenhagen University Hospital, Rigshospitalet.
Growth and Reproduction (explorative outcome) | within 2 weeks of treatment initiation.
  DNA purified from the blood samples will be analyzed for growth-factors gene polymorphism by PCR based technologies including insulin-like growth factor 1 (IGF-1), insulin-like growth factor binding protein 3 (IGFBP-3), testosterone (and tumor necrosis factor-alpha (TNF-α)) in collaboration with Department for Growth and Reproduction, Copenhagen University Hospital, Rigshospitalet.
Growth and Reproduction (explorative outcome) | 6 months after inclusion (before a treatment block)
  DNA purified from the blood samples will be analyzed for growth-factors gene polymorphism by PCR based technologies including insulin-like growth factor 1 (IGF-1), insulin-like growth factor binding protein 3 (IGFBP-3), testosterone (and tumor necrosis factor-alpha (TNF-α)) in collaboration with Department for Growth and Reproduction, Copenhagen University Hospital, Rigshospitalet.
Growth and Reproduction (explorative outcome) | 1 month after ended treatment.
  DNA purified from the blood samples will be analyzed for growth-factors gene polymorphism by PCR based technologies including insulin-like growth factor 1 (IGF-1), insulin-like growth factor binding protein 3 (IGFBP-3), testosterone (and tumor necrosis factor-alpha (TNF-α)) in collaboration with Department for Growth and Reproduction, Copenhagen University Hospital, Rigshospitalet.
Growth and Reproduction (explorative outcome) | 1 year after end of treatment.
  DNA purified from the blood samples will be analyzed for growth-factors gene polymorphism by PCR based technologies including insulin-like growth factor 1 (IGF-1), insulin-like growth factor binding protein 3 (IGFBP-3), testosterone (and tumor necrosis factor-alpha (TNF-α)) in collaboration with Department for Growth and Reproduction, Copenhagen University Hospital, Rigshospitalet.
Muscle Power: Counter Movement Jump (Rate of Force Development)(explorative outcome) | Within 2 weeks of treatment initiation (baseline)
  All counter movement jumps are carried out on a mobile force plate platform (FP4, HUR-Labs Oy, Tampere, Finland). The participant is given instructions on how to perform the CMJ correctly and is given time to familiarize with each test.
  The participant stands with both hands resting on the hips. Both hands must stay in this position during the test. The knee angle movement is standardized; participant is instructed to bend down until knees is in a 90-degree angle and immediately hereafter jumps a s high as possible in a vertical direction, landing on both feet simultaneously on the platform.
  Three attempts with a one-minute break is carried out, however the participant can try as many attempts as possible if the participant keeps showing improvements. The highest score is noted.
  Depending on tumor location, children with solid tumors may be restricted to participate in the counter movement jump.
Muscle Power: Counter Movement Jump (Rate of Force Development)(explorative outcome) | 6-months after inclusion
  All counter movement jumps are carried out on a mobile force plate platform (FP4, HUR-Labs Oy, Tampere, Finland). The participant is given instructions on how to perform the CMJ correctly and is given time to familiarize with each test.
  The participant stands with both hands resting on the hips. Both hands must stay in this position during the test. The knee angle movement is standardized; participant is instructed to bend down until knees is in a 90-degree angle and immediately hereafter jumps a s high as possible in a vertical direction, landing on both feet simultaneously on the platform.
  Three attempts with a one-minute break is carried out, however the participant can try as many attempts as possible if the participant keeps showing improvements. The highest score is noted.
  Depending on tumor location, children with solid tumors may be restricted to participate in the counter movement jump.
Muscle Power: Counter Movement Jump (Rate of Force Development)(explorative outcome) | 3-months after inclusion
  All counter movement jumps are carried out on a mobile force plate platform (FP4, HUR-Labs Oy, Tampere, Finland). The participant is given instructions on how to perform the CMJ correctly and is given time to familiarize with each test.
  The participant stands with both hands resting on the hips. Both hands must stay in this position during the test. The knee angle movement is standardized; participant is instructed to bend down until knees is in a 90-degree angle and immediately hereafter jumps a s high as possible in a vertical direction, landing on both feet simultaneously on the platform.
  Three attempts with a one-minute break is carried out, however the participant can try as many attempts as possible if the participant keeps showing improvements. The highest score is noted.
  Depending on tumor location, children with solid tumors may be restricted to participate in the counter movement jump.
Muscle Power: Counter Movement Jump (Rate of Force Development)(explorative outcome) | 1 month after ended treatment
  All counter movement jumps are carried out on a mobile force plate platform (FP4, HUR-Labs Oy, Tampere, Finland). The participant is given instructions on how to perform the CMJ correctly and is given time to familiarize with each test.
  The participant stands with both hands resting on the hips. Both hands must stay in this position during the test. The knee angle movement is standardized; participant is instructed to bend down until knees is in a 90-degree angle and immediately hereafter jumps a s high as possible in a vertical direction, landing on both feet simultaneously on the platform.
  Three attempts with a one-minute break is carried out, however the participant can try as many attempts as possible if the participant keeps showing improvements. The highest score is noted.
  Depending on tumor location, children with solid tumors may be restricted to participate in the counter movement jump.
Muscle Power: Counter Movement Jump (Rate of Force Development)(explorative outcome) | 1 year after ended treatment
  All counter movement jumps are carried out on a mobile force plate platform (FP4, HUR-Labs Oy, Tampere, Finland). The participant is given instructions on how to perform the CMJ correctly and is given time to familiarize with each test.
  The participant stands with both hands resting on the hips. Both hands must stay in this position during the test. The knee angle movement is standardized; participant is instructed to bend down until knees is in a 90-degree angle and immediately hereafter jumps a s high as possible in a vertical direction, landing on both feet simultaneously on the platform.
  Three attempts with a one-minute break is carried out, however the participant can try as many attempts as possible if the participant keeps showing improvements. The highest score is noted.
  Depending on tumor location, children with solid tumors may be restricted to participate in the counter movement jump.
Neuropathy - Ped-mTNS (explorative outcome) | Within 2 weeks of treatment initiation (baseline)
  Neuropathy is evaluated using the Pediatric Modified Total Neuropathy Score (Ped-mTNS)(72). This validated instrument captures impairment-level information on the function of the peripheral nervous system and includes questions on sensory, motor, and autonomic symptoms; examination of light touch, pin, and vibration perception; muscle strength of distal musculature; and deep tendon reflexes.
Neuropathy - Ped-mTNS (explorative outcome) | 3-months after inclusion
  Neuropathy is evaluated using the Pediatric Modified Total Neuropathy Score (Ped-mTNS)(72). This validated instrument captures impairment-level information on the function of the peripheral nervous system and includes questions on sensory, motor, and autonomic symptoms; examination of light touch, pin, and vibration perception; muscle strength of distal musculature; and deep tendon reflexes.
Neuropathy - Ped-mTNS (explorative outcome) | 6-months after inclusion
  Neuropathy is evaluated using the Pediatric Modified Total Neuropathy Score (Ped-mTNS)(72). This validated instrument captures impairment-level information on the function of the peripheral nervous system and includes questions on sensory, motor, and autonomic symptoms; examination of light touch, pin, and vibration perception; muscle strength of distal musculature; and deep tendon reflexes.
Neuropathy - Ped-mTNS (explorative outcome) | one month after ended treatment
  Neuropathy is evaluated using the Pediatric Modified Total Neuropathy Score (Ped-mTNS)(72). This validated instrument captures impairment-level information on the function of the peripheral nervous system and includes questions on sensory, motor, and autonomic symptoms; examination of light touch, pin, and vibration perception; muscle strength of distal musculature; and deep tendon reflexes.
Neuropathy - Ped-mTNS (explorative outcome) | 1 year after ended treatment
  Neuropathy is evaluated using the Pediatric Modified Total Neuropathy Score (Ped-mTNS)(72). This validated instrument captures impairment-level information on the function of the peripheral nervous system and includes questions on sensory, motor, and autonomic symptoms; examination of light touch, pin, and vibration perception; muscle strength of distal musculature; and deep tendon reflexes.
Physio- and occupational therapy treatments (explorative outcome) | measured 6 months after inclusion
  Total number physiotherapy and occupational therapy treaments (days) will be drawn from the participants medical records.
Physio- and occupational therapy treatments (explorative outcome) | 1 month after ended treatment
  Total number physiotherapy and occupational therapy treaments (days) will be drawn from the participants medical records.
Physio- and occupational therapy treatments (explorative outcome) | 1 year after ended treatment
  Total number physiotherapy and occupational therapy treaments (days) will be drawn from the participants medical records.
General Physical Acivity: Young Children (6-7 years), Children (8-12 years), Teens (13-18 years) Self-Report and Parent Proxy-Report (explorative outcome) | Within 2 weeks of treatment initiation.
  An validated questionnaire used in the UNGkan and HEIA project will be used to assess self-reported physical activity, physical function, sedentary time, screen time, diet habits, active transportation behavior, physical education participation, perceived barriers/facilitators to physical activity, health-related behaviors. The questionnaire contains four versions targeted either children (<14 years) or youth (>14 years) and the parents guardians to each of these subgroups. The questionnaire contains 35 items for the child/youth report and 18 items for the parent proxy report for both groups.
General Physical Acivity: Young Children (6-7 years), Children (8-12 years), Teens (13-18 years) Self-Report and Parent Proxy-Report: (explorative outcome) | 6-months after inclusion.
  An validated questionnaire used in the UNGkan and HEIA project will be used to assess self-reported physical activity, physical function, sedentary time, screen time, diet habits, active transportation behavior, physical education participation, perceived barriers/facilitators to physical activity, health-related behaviors. The questionnaire contains four versions targeted either children (<14 years) or youth (>14 years) and the parents guardians to each of these subgroups. The questionnaire contains 35 items for the child/youth report and 18 items for the parent proxy report for both groups.
General Physical Acivity: Young Children (6-7 years), Children (8-12 years), Teens (13-18 years) Self-Report and Parent Proxy-Report (explorative outcome) | 1 month after ended treatment.
  An validated questionnaire used in the UNGkan and HEIA project will be used to assess self-reported physical activity, physical function, sedentary time, screen time, diet habits, active transportation behavior, physical education participation, perceived barriers/facilitators to physical activity, health-related behaviors. The questionnaire contains four versions targeted either children (<14 years) or youth (>14 years) and the parents guardians to each of these subgroups. The questionnaire contains 35 items for the child/youth report and 18 items for the parent proxy report for both groups.
General Physical Acivity: Young Children (6-7 years), Children (8-12 years), Teens (13-18 years) Self-Report and Parent Proxy-Report (explorative outcome) | 1 year after ended treatment.
  An validated questionnaire used in the UNGkan and HEIA project will be used to assess self-reported physical activity, physical function, sedentary time, screen time, diet habits, active transportation behavior, physical education participation, perceived barriers/facilitators to physical activity, health-related behaviors. The questionnaire contains four versions targeted either children (<14 years) or youth (>14 years) and the parents guardians to each of these subgroups. The questionnaire contains 35 items for the child/youth report and 18 items for the parent proxy report for both groups.
The PedsQL 3.0 Cancer Scale: Young Child, Children, Teens Self-Report and Parent Proxy-Report | Within 2 weeks of treatment initiation.
  The PedsQL 3.0 Cancer Module instrument encompasses eight subscales: (1) pain and hurt, (2) nausea, (3) procedural anxiety, (4) treatment anxiety, (5) worry, (6) cognitive problems, (7) perceived physical appearance, and (8) communication
The PedsQL 3.0 Cancer Scale: Young Child, Children, Teens Self-Report and Parent Proxy-Report (explorative outcome) | 6 months after inclusion
  The PedsQL 3.0 Cancer Module instrument encompasses eight subscales: (1) pain and hurt, (2) nausea, (3) procedural anxiety, (4) treatment anxiety, (5) worry, (6) cognitive problems, (7) perceived physical appearance, and (8) communication
PedsQL Multidimensional Fatigue Scale: Young Child, Children, Teens Self-Report and Parent Proxy-Report (explorative outcome) | Within 2 weeks of treatment initiation.
  Composed og 18 items, the PedsQL Multidimensional Fatigue Scale possesses three subscales: general fatigue, sleep and rest fatigue, and cognitive fatigue.
PedsQL Multidimensional Fatigue Scale: Young Child, Children, Teens Self-Report and Parent Proxy-Report (explorative outcome) | 6 months after inclusion.
  Composed og 18 items, the PedsQL Multidimensional Fatigue Scale possesses three subscales: general fatigue, sleep and rest fatigue, and cognitive fatigue.
PedsQL Multidimensional Fatigue Scale: Young Child, Children, Teens Self-Report and Parent Proxy-Report (explorative outcome) | 1 month after ended treatment.
  Composed og 18 items, the PedsQL Multidimensional Fatigue Scale possesses three subscales: general fatigue, sleep and rest fatigue, and cognitive fatigue.
PedsQL Multidimensional Fatigue Scale: Young Child, Children, Teens Self-Report and Parent Proxy-Report (explorative outcome) | 1 year after end of treatment.
  Composed og 18 items, the PedsQL Multidimensional Fatigue Scale possesses three subscales: general fatigue, sleep and rest fatigue, and cognitive fatigue.
Self-Efficacy for Exercise scale (SEE-DK) (explorative outcome) | monthly, up to 6 months after inclusion
  Self-efficacy for exercise is measured using the Danish version of the SEE scale. This scale contains nine-items concerning nine different potential barriers (weather, activity being tedious, pain, loneliness, disliking the activity, irrelevance, fatigue, stress, sadness) to perform physical exercise.
Modified Clinical Test of Sensory Interaction in Balance (explorative outcome) | Within 2 weeks of treatment initiation (baseline)
  This four-condition test is designed to assess how well an individual is using sensory inputs to maintain balance when one or more sensory systems are compromised. In condition one, all sensory systems (i.e., vision, somatosensory, and vestibular) are available for maintaining balance. In condition two, vision has been removed and the participant must rely on the somatosensory and vestibular systems to balance. In condition three, the somatosensory system has been compromised and the participant must use vision and the vestibular system to balance. In condition four, vision has been removed and the somatosensory system has been compromised.
  Each trial is timed using a stopwatch. The trial is over when (a) the participant opens his/her eyes in an eyes closed condition, (b) raises arms from sides, (c) loses balance and requires manual assistance to prevent a fall or (d) maintains balance for 30 seconds.
Modified Clinical Test of Sensory Interaction in Balance (explorative outcome) | 3-months after inclusion
  This four-condition test is designed to assess how well an individual is using sensory inputs to maintain balance when one or more sensory systems are compromised. In condition one, all sensory systems (i.e., vision, somatosensory, and vestibular) are available for maintaining balance. In condition two, vision has been removed and the participant must rely on the somatosensory and vestibular systems to balance. In condition three, the somatosensory system has been compromised and the participant must use vision and the vestibular system to balance. In condition four, vision has been removed and the somatosensory system has been compromised.
  Each trial is timed using a stopwatch. The trial is over when (a) the participant opens his/her eyes in an eyes closed condition, (b) raises arms from sides, (c) loses balance and requires manual assistance to prevent a fall or (d) maintains balance for 30 seconds.
Modified Clinical Test of Sensory Interaction in Balance (explorative outcome) | 6-months after inclusion
  This four-condition test is designed to assess how well an individual is using sensory inputs to maintain balance when one or more sensory systems are compromised. In condition one, all sensory systems (i.e., vision, somatosensory, and vestibular) are available for maintaining balance. In condition two, vision has been removed and the participant must rely on the somatosensory and vestibular systems to balance. In condition three, the somatosensory system has been compromised and the participant must use vision and the vestibular system to balance. In condition four, vision has been removed and the somatosensory system has been compromised.
  Each trial is timed using a stopwatch. The trial is over when (a) the participant opens his/her eyes in an eyes closed condition, (b) raises arms from sides, (c) loses balance and requires manual assistance to prevent a fall or (d) maintains balance for 30 seconds.
Modified Clinical Test of Sensory Interaction in Balance (explorative outcome) | 1 month after ended treatment
  This four-condition test is designed to assess how well an individual is using sensory inputs to maintain balance when one or more sensory systems are compromised. In condition one, all sensory systems (i.e., vision, somatosensory, and vestibular) are available for maintaining balance. In condition two, vision has been removed and the participant must rely on the somatosensory and vestibular systems to balance. In condition three, the somatosensory system has been compromised and the participant must use vision and the vestibular system to balance. In condition four, vision has been removed and the somatosensory system has been compromised.
  Each trial is timed using a stopwatch. The trial is over when (a) the participant opens his/her eyes in an eyes closed condition, (b) raises arms from sides, (c) loses balance and requires manual assistance to prevent a fall or (d) maintains balance for 30 seconds.
Modified Clinical Test of Sensory Interaction in Balance (explorative outcome) | 1 year after ended treatment
  This four-condition test is designed to assess how well an individual is using sensory inputs to maintain balance when one or more sensory systems are compromised. In condition one, all sensory systems (i.e., vision, somatosensory, and vestibular) are available for maintaining balance. In condition two, vision has been removed and the participant must rely on the somatosensory and vestibular systems to balance. In condition three, the somatosensory system has been compromised and the participant must use vision and the vestibular system to balance. In condition four, vision has been removed and the somatosensory system has been compromised.
  Each trial is timed using a stopwatch. The trial is over when (a) the participant opens his/her eyes in an eyes closed condition, (b) raises arms from sides, (c) loses balance and requires manual assistance to prevent a fall or (d) maintains balance for 30 seconds.
Facilitators and Barriers to Physical Activity, semi-structured in-depth interviews (explorative outcome) | within 6-months after treatment initiation
  We will interview at least 20 children and their parents from the intervention and control group purposely sampled to represent children with high and low physical activity levels, from all centers, representatives for age, diagnosis and sex.
Physical Activity behaviour (explorative outcome) | 1 year after ended treatment.
  Physical activity and sedentary time are assessed by accelerometers worn for 7 days during and after treatment. The accelerometers (ActiGraph™ model GT3X+, ActiGraph LLC, Pensacola FL, USA) measures accelerations of ±6 G. The sample rate will be set to measure raw signals at 100 Hz, translated into metabolic energy equivalents of light, moderate and vigorous physical activity and sedentary time.
Physical Activity behaviour (explorative outcome) | 1 month after ended treatment.
  Physical activity and sedentary time are assessed by accelerometers worn for 7 days during and after treatment. The accelerometers (ActiGraph™ model GT3X+, ActiGraph LLC, Pensacola FL, USA) measures accelerations of ±6 G. The sample rate will be set to measure raw signals at 100 Hz, translated into metabolic energy equivalents of light, moderate and vigorous physical activity and sedentary time.
Physical Activity behaviour (explorative outcome) | 6-months after inclusion (primary endpoint).
  Physical activity and sedentary time are assessed by accelerometers worn for 7 days during and after treatment. The accelerometers (ActiGraph™ model GT3X+, ActiGraph LLC, Pensacola FL, USA) measures accelerations of ±6 G. The sample rate will be set to measure raw signals at 100 Hz, translated into metabolic energy equivalents of light, moderate and vigorous physical activity and sedentary time.
Physical Activity behaviour (explorative outcome) | 3-months after inclusion
  Physical activity and sedentary time are assessed by accelerometers worn for 7 days during and after treatment. The accelerometers (ActiGraph™ model GT3X+, ActiGraph LLC, Pensacola FL, USA) measures accelerations of ±6 G. The sample rate will be set to measure raw signals at 100 Hz, translated into metabolic energy equivalents of light, moderate and vigorous physical activity and sedentary time.
Physical Activity behaviour (explorative outcome) | Within 2 weeks of treatment initiation
  Physical activity and sedentary time are assessed by accelerometers worn for 7 days during and after treatment. The accelerometers (ActiGraph™ model GT3X+, ActiGraph LLC, Pensacola FL, USA) measures accelerations of ±6 G. The sample rate will be set to measure raw signals at 100 Hz, translated into metabolic energy equivalents of light, moderate and vigorous physical activity and sedentary time.
Risk factors of metabolic syndrome: Body Mass Index | within 2 weeks of treatment initiation
  Weight and Height is combined to report BMI in kg/m^2
Risk factors of metabolic syndrome: Body Mass Index | 6 months after inclusion (before a treatment block)
  Weight and Height is combined to report BMI in kg/m^2
Risk factors of metabolic syndrome: Body Mass Index | 1 month after ended treatment
  Weight and Height is combined to report BMI in kg/m^2
Risk factors of metabolic syndrome: Body Mass Index | 1 year after end of treatment (primary endpoint)
  Weight and Height is combined to report BMI in kg/m^2
Risk factors of metabolic syndrome: total cholesterol and low-density lipoprotein (LDL) cholesterol | within 2 weeks of treatment initiation
  Blood samples is reported in mmol/L
Risk factors of metabolic syndrome: total cholesterol and low-density lipoprotein (LDL) cholesterol | 6 months after inclusion (before a treatment block)
  Blood samples is reported in mmol/L
Risk factors of metabolic syndrome: total cholesterol and low-density lipoprotein (LDL) cholesterol | 1 month after ended treatment
  Blood samples is reported in mmol/L
Risk factors of metabolic syndrome: total cholesterol and low-density lipoprotein (LDL) cholesterol | 1 year after end of treatment (primary endpoint)
  Blood samples is reported in mmol/L
Risk factors of metabolic syndrome: Oral Glucose Tolerance Test | within 2 weeks of treatment initiation
  An Oral Glucose Tolerance Test is performed in the morning following an overnight fast initiated at 10:00 pm the previous evening. Participants will receive 1.75 g/kg of dextrose (maximum of 75 g). Blood will be sampled for serum insulin and plasma glucose at fasting and at 30, 60, 90 and 120 minutes after dextrose administration. Insulin concentrations is determined using an immunochemiluminometric assay. The insulin assay uses a monoclonal anti-insulin antibody and was run on an Immulite2000 machine (Diagnostic Product Corporation, Los Angeles, California).
Risk factors of metabolic syndrome: Oral Glucose Tolerance Test | 6 months after inclusion (before a treatment block)
  An Oral Glucose Tolerance Test is performed in the morning following an overnight fast initiated at 10:00 pm the previous evening. Participants will receive 1.75 g/kg of dextrose (maximum of 75 g). Blood will be sampled for serum insulin and plasma glucose at fasting and at 30, 60, 90 and 120 minutes after dextrose administration. Insulin concentrations is determined using an immunochemiluminometric assay. The insulin assay uses a monoclonal anti-insulin antibody and was run on an Immulite2000 machine (Diagnostic Product Corporation, Los Angeles, California).
Risk factors of metabolic syndrome: Oral Glucose Tolerance Test | 1 month after ended treatment
  An Oral Glucose Tolerance Test is performed in the morning following an overnight fast initiated at 10:00 pm the previous evening. Participants will receive 1.75 g/kg of dextrose (maximum of 75 g). Blood will be sampled for serum insulin and plasma glucose at fasting and at 30, 60, 90 and 120 minutes after dextrose administration. Insulin concentrations is determined using an immunochemiluminometric assay. The insulin assay uses a monoclonal anti-insulin antibody and was run on an Immulite2000 machine (Diagnostic Product Corporation, Los Angeles, California).
Risk factors of metabolic syndrome: Oral Glucose Tolerance Test | 1 year after end of treatment (primary endpoint)
  An Oral Glucose Tolerance Test is performed in the morning following an overnight fast initiated at 10:00 pm the previous evening. Participants will receive 1.75 g/kg of dextrose (maximum of 75 g). Blood will be sampled for serum insulin and plasma glucose at fasting and at 30, 60, 90 and 120 minutes after dextrose administration. Insulin concentrations is determined using an immunochemiluminometric assay. The insulin assay uses a monoclonal anti-insulin antibody and was run on an Immulite2000 machine (Diagnostic Product Corporation, Los Angeles, California).
Risk factors of metabolic syndrome: hip circumference | within 2 weeks of treatment initiation
  Hip circumference (in CM) at a level parallel to the floor, at the largest circumference of the buttocks following standards described by the World Health Organization. Metabolic syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Risk factors of metabolic syndrome: hip circumference | 6 months after inclusion (before a treatment block)
  Hip circumference (in CM) at a level parallel to the floor, at the largest circumference of the buttocks following standards described by the World Health Organization. Metabolic syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Risk factors of metabolic syndrome: hip circumference | 1 month after ended treatment
  Hip circumference (in CM) at a level parallel to the floor, at the largest circumference of the buttocks following standards described by the World Health Organization. Metabolic syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).
Risk factors of metabolic syndrome: hip circumference | 1 year after end of treatment (primary endpoint)
  Hip circumference (in CM) at a level parallel to the floor, at the largest circumference of the buttocks following standards described by the World Health Organization. Metabolic syndrome is based on age-based criterias defined by the International Diabetes Foundation (3).

CONTACTS AND LOCATIONS:
Overall Officials: Hanne B. Larsen, As. Prof, Principal Investigator — Rigshospitalet, Denmark
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thorsteinsson T, Helms AS, Adamsen L, Andersen LB, Andersen KV, Christensen KB, Hasle H, Heilmann C, Hejgaard N, Johansen C, Madsen M, Madsen SA, Simovska V, Strange B, Thing LF, Wehner PS, Schmiegelow K, Larsen HB. Study protocol: Rehabilitation including Social and Physical activity and Education in Children and Teenagers with Cancer (RESPECT). BMC Cancer. 2013 Nov 14;13:544. doi: 10.1186/1471-2407-13-544. PMID 24229362
- [Background] Fiuza-Luces C, Padilla JR, Soares-Miranda L, Santana-Sosa E, Quiroga JV, Santos-Lozano A, Pareja-Galeano H, Sanchis-Gomar F, Lorenzo-Gonzalez R, Verde Z, Lopez-Mojares LM, Lassaletta A, Fleck SJ, Perez M, Perez-Martinez A, Lucia A. Exercise Intervention in Pediatric Patients with Solid Tumors: The Physical Activity in Pediatric Cancer Trial. Med Sci Sports Exerc. 2017 Feb;49(2):223-230. doi: 10.1249/MSS.0000000000001094. PMID 27631396
- [Background] Zimmet P, Alberti KG, Kaufman F, Tajima N, Silink M, Arslanian S, Wong G, Bennett P, Shaw J, Caprio S; IDF Consensus Group. The metabolic syndrome in children and adolescents - an IDF consensus report. Pediatr Diabetes. 2007 Oct;8(5):299-306. doi: 10.1111/j.1399-5448.2007.00271.x. No abstract available. PMID 17850473
- [Derived] Schmidt-Andersen P, Fridh MK, Muller KG, Anna Pouplier, Hjalgrim LL, Faigenbaum AD, Schmiegelow K, Hasle H, Lykkedegn S, Zhang H, Christensen J, Larsen HB. Integrative Neuromuscular Training in Adolescents and Children Treated for Cancer (INTERACT): Study Protocol for a Multicenter, Two-Arm Parallel-Group Randomized Controlled Superiority Trial. Front Pediatr. 2022 Mar 14;10:833850. doi: 10.3389/fped.2022.833850. eCollection 2022. PMID 35359909